CLINICAL TRIAL: NCT03626415
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE STUDY TO COMPARE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-04965842 IN ADULT SUBJECTS WITH MILD AND MODERATE HEPATIC IMPAIRMENT RELATIVE TO SUBJECTS WITH NORMAL HEPATIC FUNCTION
Brief Title: A Hepatic Impairment Study for PF-04965842.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7451020
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: Recruitment for subjects with moderate and mild hepatic impairment (Cohorts 1 and 2) will initiate first and these subjects will be enrolled in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-04965842 (Experimental): PF 04965842 is an orally bioavailable small molecule that selectively inhibits JAK1.
  Interventions: Drug: PF-04965842

INTERVENTIONS:
Drug: PF-04965842 — PF 04965842 is an orally bioavailable small molecule that selectively inhibits JAK1.

SUMMARY:
This is a Phase 1 non randomized, open label, single dose, parallel cohort study to investigate the effect of hepatic impairment on the PK, safety and tolerability of PF 04965842.

DETAILED DESCRIPTION:
A minimum of 24 subjects with normal, mild or moderate hepatic function will be enrolled into the study, with approximately 8 subjects in each cohort. The Child Pugh classification score will be utilized to assess entry criteria and to assign subjects into the appropriate hepatic impairment group. For individual subjects, the total maximum duration of study participation from the Screening visit to the end of clinical research unit (CRU) stay is approximately 31 days and approximately 63 days from the Screening visit to the Follow up contact.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 pounds).
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Additional Inclusion Criteria for subjects with hepatic impairment:

* Satisfy the criteria for Class A or Class B of the Child Pugh classification (mild: Child Pugh Scores 5 to 6 points, and moderate: Child Pugh Scores 7 to 9 points), within 14 days of investigational product administration.
* A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography scan, or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Subjects with clinically significant infections within the past 3 months (for example, those requiring hospitalization, or as judged by the Investigator), evidence of any infection (including influenza) within the past 7 days, history of disseminated herpes simplex infection or recurrent (>1 episode) or disseminated herpes zoster.
* Subjects with a malignancy or with a history of malignancy, with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Additional exclusion criteria for subjects with hepatic impairment:

* Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy (defined as less than 1 year).
* Subjects who have previously had a transplanted kidney, liver, or heart.
* At Screening, persistent severe, uncontrolled hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Clinical Research, LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- [Derived] Wang EQ, Le V, O'Gorman M, Tripathy S, Dowty ME, Wang L, Malhotra BK. Effects of Hepatic Impairment on the Pharmacokinetics of Abrocitinib and Its Metabolites. J Clin Pharmacol. 2021 Oct;61(10):1311-1323. doi: 10.1002/jcph.1858. Epub 2021 Apr 17. PMID 33749838
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451020

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04965842 (Normal Hepatic Function Cohort): Participants with normal hepatic function were enrolled in this cohort. Participants received a single oral dose of PF-04965842 200 mg.
- PF-04965842 (Mild Hepatic Impairment Cohort): Participants with Child-Pugh scores of 5 to 6 points were enrolled in this cohort. Participants received a single oral dose of PF-04965842 200 mg.
- PF-04965842 (Moderate Hepatic Impairment Cohort): Participants with Child-Pugh scores of 7 to 9 points were enrolled in this cohort. Participants received a single oral dose of PF-04965842 200 mg.
Period: Overall Study
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (5.86) | 57.9 (4.19) | 58.6 (8.21) | 58.3 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 5 | 5 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 5
  White | 7 | 4 | 7 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-04965842
Description: Cmax is maximum plasma concentration. It was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72 hours post-dose in each cohort
Population: The pharmacokinetic concentration population was defined as all participants who received 1 dose of PF-04965842 and in whom at least 1 plasma concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter (ng/mL) | 1352 (44) | 1276 (41) | 1426 (63)
Statistical Analysis 1: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Mild Hepatic Impairment Cohort); Mild Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Mean = 94.40, 90% CI 2-sided [62.96 to 141.55]
Statistical Analysis 2: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Moderate Hepatic Impairment Cohort); Moderate Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adusted Geometric Means = 105.53, 90% CI 2-sided [70.38 to 158.24]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) for PF-04965842
Description: AUCinf is area under the concentration-time curve (AUC) from time 0 (pre-dose) extrapolated to infinite time.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72 hours post-dose in each cohort
Population: The pharmacokinetic parameter analysis population was defined as all participants dosed who had at least 1 of the pharmocokinetics parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
nanogram*hour per milliliter (ng*hr/mL) | 5587 (74) | 7449 (29) | 8603 (55)
Statistical Analysis 1: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Mild Hepatic Impairment Cohort); Mild Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 133.33, 90% CI 2-sided [86.17 to 206.28]
Statistical Analysis 2: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Moderate Hepatic Impairment Cohort); Moderate Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Mean = 153.99, 90% CI 2-sided [99.52 to 238.25]

3. Post Hoc Outcome: Unbound Cmax (Cmax,u) for Active Moiety
Description: Cmax,u is unbound Cmax. The active moiety is comprised of parent drug PF-04965842, active metabolites PF-06471658 and PF-07055087.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72 hours post-dose in each cohort
Population: The pharmacokinetic parameter analysis population was defined as all participants dosed who had at least 1 of the pharmocokinetic parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
nanomolar (nM) | 2390 (20) | 1815 (36) | 2011 (41)
Statistical Analysis 1: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Mild Hepatic Impairment Cohort); Mild Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 75.94, 90% CI 2-sided [57.39 to 100.47]
Statistical Analysis 2: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Moderate Hepatic Impairment Cohort); Moderate Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 84.14, 90% CI 2-sided [63.59 to 111.33]

4. Post Hoc Outcome: Unbound AUCinf (AUCinf,u) for Active Moiety
Description: AUCinf,u is unbound AUCinf. The active moiety is comprised of parent drug PF-04965842, active metabolites PF-06471658 and PF-07055087.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72 hours post-dose in each cohort
Population: The analysis population was defined as all participants contributing to the summary statistics for AUCinf,u.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar*hour (nM*hr)
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 7 | 8 | 8
nanomolar*hour (nM*hr) | 12010 (40) | 11500 (24) | 13790 (30)
Statistical Analysis 1: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Mild Hepatic Impairment Cohort); Mild Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 95.74, 90% CI 2-sided [72.71 to 126.08]
Statistical Analysis 2: Comparison: PF-04965842 (Normal Hepatic Function Cohort) vs PF-04965842 (Moderate Hepatic Impairment Cohort); Moderate Hepatic Impairment (Test) versus Normal Hepatic Function (Reference); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 114.82, 90% CI 2-sided [87.19 to 151.20]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) for PF-04965842
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent adverse events (TEAEs) were those with initial onset or increasing in severity between the first dose of investigational product and up to 36 days post-dose.
Time Frame: From screening (within 28 days prior to Day 1) till up to 36 days post-dose, the total maximum duration was approximately 63 days for individual participants.
Population: All participants who received PF-04965842 were included in the safety analyses.
Measure: Number; unit: Participants
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
Participants
  AEs (all causalities) | 2 | 3 | 0
  AEs (treatment related) | 1 | 3 | 0

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included tests that were performed under the categories of hematology, chemistry, urinalysis, other, and additional tests needed for Hy's law.
Time Frame: Screening (within 28 days prior to Day 1), Day -1, 2, 24, 72 hours post-dose.
Population: All participants who received PF-04965842 were included in the safety analyses.
Measure: Number; unit: Participants
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
Participants | 4 | 7 | 8

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings of Potential Clinical Importance for PF-04965842
Description: 12-Lead ECGs were collected after the participants rested quietly for at least 10 minutes in a supine position. Clinical significance of ECG recordings was determined at the investigator's discretion.
Time Frame: Screening (within 28 days prior to Day 1), Day -1, 2, 72 hours post-dose.
Population: All participants who received PF-04965842 were included in the safety analyses.
Measure: Number; unit: Participants
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Vital Sign Findings of Potential Clinical Importance for PF-04965842
Description: Vital signs (pulse rate, systolic and diastolic blood pressure) were obtained with participant following at least 5 minutes of supine rest. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Screening (within 28 days prior to Day 1), 0 (pre-dose), and 72 hours post-dose.
Population: All participants who received PF-04965842 were included in the safety analyses.
Measure: Number; unit: Participants
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening (within 28 days prior to Day 1) till up to 36 days post-dose, the total maximum duration was approximately 63 days for individual participants.
Arm/Group | PF-04965842 (Normal Hepatic Function Cohort) | PF-04965842 (Mild Hepatic Impairment Cohort) | PF-04965842 (Moderate Hepatic Impairment Cohort)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 3/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 (Normal Hepatic Function Cohort) (N=8) | PF-04965842 (Mild Hepatic Impairment Cohort) (N=8) | PF-04965842 (Moderate Hepatic Impairment Cohort) (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03626415/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03626415/SAP_001.pdf